CLINICAL TRIAL: NCT00665210
Title: Photo-manipulation of Digital Radiographs and Digitized Templates as a Method for Preoperative Sizing of Total Hip Arthroplasties
Brief Title: Digital Sizing for Orthopaedic Hip Implants
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2007-511
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Last update posted 2011-10-26 (Estimated); Status verified 2011-10

CONDITIONS: Hip Arthritis
Keywords: hip arthritis; implant sizing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Hip implants come in different sizes. Currently, surgeons predict the implant size that will be needed using an analogue method whereby photos of the implant sizes are overlaid on the x-rays. In this study, we propose to use a digital, computerized method of templating which we expect will be more accurate than the overlay method.

ELIGIBILITY:
Inclusion Criteria:

* Patients booked for primary total hip arthroplasty with non-cemented prosthesis.
* No previous surgery/fractures to acetabulum or femur or hip.
* No gross bony abnormality except for osteoarthritis and avascular necrosis.

Exclusion Criteria:

* Cancer or tumor suspected, morbid obesity, revision, previous acetabular/femur/hip surgery, gross bony deformity, calibration bar not completely pictured on radiograph, unsuccessful surgery fracture/cancer/cemented prosthesis used.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients booked for primary total hip arthroplasty with non-cemented prosthesis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-10

CONTACTS AND LOCATIONS:
Overall Officials: Peter Thurston, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- OHRI, Ottawa, Ontario, Canada